CLINICAL TRIAL: NCT03119272
Title: Microbiome-mediated Weight, Anxiety, and Stress Dysregulation in Anorexia Nervosa
Acronym: Microbiome
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 15-2133; 1R01MH105684-01A1 (NIH)
Record Dates: First submitted 2016-04-04; First posted 2017-04-18 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Anorexia Nervosa Patients: Inpatient population at Eating Disorders Unit (EDU) at the University of North Carolina Neurosciences Hospital. Recruited upon intake into the unit.
- Age and Sex Matched Healthy Controls: University of North Carolina Psychiatry email listserv.

SUMMARY:
The purpose of this research study is to analyze the microorganisms residing in the gut of patients with anorexia nervosa. Research has begun to link changes in the intestinal microbiota with diseases such as inflammatory bowel disease (IBS), asthma, and obesity, but although some studies have investigated the intestinal microbiota in overweight/obese individuals, very little is known about the intestinal microbiota in underweight individuals. The investigators aim to identify the enteric bacterial groups associated with adiposity, BMI, anxiety, and stress in patients with anorexia nervosa.

DETAILED DESCRIPTION:
Anorexia nervosa (AN), a psychiatric disorder characterized by extreme weight dysregulation commonly presents with comorbid anxiety. Therapeutic renourishment in AN is based primarily on clinical opinion and guidelines, with a weak evidence base. Compelling data implicate the intestinal microbiota in the regulation of adiposity and behavior, providing a strong rationale for exploring the role of this complex microbial community in the emergence and maintenance of, and recovery from AN. The overarching goal is to understand the precise mechanism(s) by which intestinal bacteria contribute to dysregulation of adiposity, BMI, anxiety, and stress in patients with AN. The investigators hypothesize that intestinal microbiotas that arise from prolonged starvation contribute to increases in adiposity upon refeeding and to persistently elevated anxiety and stress in individuals with AN. To test the hypothesis the investigators propose 3 specific aims. In aim 1, the investigators will identify the enteric bacterial groups associated with adiposity, BMI, anxiety, and stress in AN patients. The investigators will characterize the intestinal microbiota in acutely low weight AN patients (T1), in the same patients following weight restoration (T2), and in healthy controls (HC) via high throughput sequencing of the 16S rRNA gene.

The investigators will compare the abundances of specific enteric taxa with adiposity, BMI and behavior (anxiety and stress) in this study population. In aim 2, The investigators will characterize the functional impact of the intestinal microbiota of AN patients on adiposity and BMI when transplanted into germ free (GF) mice. The investigators will transplant uncultured microbiotas from AN patients (at T1 and T2) and HC into GF mice and assess the impact of enteric microbes on adiposity. In aim 3, the investigators will characterize the functional impact of the intestinal microbiota of AN patients on anxiety and stress, and molecular biomarkers of these behaviors, when transplanted into GF mice. The investigators will transplant uncultured microbiotas from T1 AN patients and HC into GF mice and assess the impact of enteric microbes on anxiety and stress. GF mice gavaged with sterile phosphate buffer saline will be used as controls in aims 2 and 3. The proposed science is significant in pioneering the combination of large scale 16S rRNA gene sequencing-based studies of intestinal microbiotas in AN with exploration of their functional influence on adiposity and behavioral traits associated with AN. The results will provide direction on how best to test adjunct interventions for AN with pre-, pro-, anti-, or syn-biotics to enhance current approaches to therapeutic weight restoration and improve treatment outcome. The science is highly innovative as it will investigate an entirely novel factor in AN, the intestinal microbiota, and use a novel approach to identify enteric microbes that impact adiposity and behavior in this devastating illness. Additionally, the investigators will hope to study an entirely novel factor (namely, the intestinal microbiota) as a contributor to the underlying pathophysiology of AN.

ELIGIBILITY:
Inclusion Criteria:

* Anorexia nervosa patient receiving treatment

Exclusion Criteria:

* history of gastrointestinal tract surgery
* history of inflammatory bowel diseases (IBD)
* history of irritable bowel syndrome (IBS)
* history of celiac disease
* history of any other diagnosis that could explain chronic or recurring bowel symptoms
* treatment in the last two months with antibiotics, non-steroid anti-inflammatory agents, or steroids.
* eating disorders or other major psychiatric or medical issue (for healthy controls).

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Inpatient population at Eating Disorders Unit (EDU) at UNC hospitals. Healthy controls pooled through UNC listserv.
Sampling Method: Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Perfect total fat as it relates to each taxa (percentage abundance from phylum to the genus level) and their association with weight. | 18 Months
  The composition and diversity of the intestinal microbiota will be characterized and correlated with adiposity. The researchers will use a DXA scan to measure this.

SECONDARY OUTCOMES:
Anxiety level (as measured by the State-Trait Anxiety Inventory) as it relates to each taxa (percentage abundance from phylum to the genus level). | 18 Months
  The composition and diversity of the intestinal microbiota will be characterized and correlated with anxiety measures.The enteric bacterial groups will be measured via percentage abundance from phylum to the genus level. Anxiety will be measured by the State-Trait Anxiety Inventory (STAI). The STAI questionnaire consists of 40 questions with 20 items allocated to each of the State Anxiety and Trait Anxiety subscales. The scores for each subtest range from 20 to 80, with higher scores indicating higher levels of anxiety.
Stress level (as measured by the Perceived Stress Scale) as it relates to taxa (percentage abundance from phylum to the genus level). | 18 Months
  The composition and diversity of the intestinal microbiota will be characterized and correlated with anxiety and stress measures.The enteric bacterial groups will be measured via percentage abundance from phylum to the genus level. Stress will be measured by the Perceived Stress Scale (PSS). The "Perceived Stress Scale" measures the overall level of stress. This instrument contains 10 items accessing overall appraisals of stress in the past month. The scale refers to the caregiver. Minimum score (best value)=0. Maximum score (worst value)=40. Higher values represent a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Carroll, PhD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Reed KK, Bulik-Sullivan EC, Qian Y, Javorsky E, Tarantino LM, Fodor AA, Steffen KJ, Wonderlich SA, Mehler PS, Bulik CM, Carroll IM. Using Bomb Calorimetry to Investigate Intestinal Energy Harvest in Anorexia Nervosa: Preliminary Findings on Stool Calorie Loss. Int J Eat Disord. 2025 Feb;58(2):440-445. doi: 10.1002/eat.24331. Epub 2024 Nov 21. PMID 39569450